CLINICAL TRIAL: NCT02982408
Title: Can Exercise Training Revert and/or Minimize the Deleterious Cardiometabolic Effects of Carbohydrate Overfeeding in Individuals With and Without Increased Risk of Type 2 Diabetes?
Brief Title: Impact of Overfeeding and Following Exercise Training in Individuals With and Without Increased Risk of Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Novo Nordisk A/S (Industry); Augustinus Fonden (Other)
Responsible Party: Principal Investigator, Charlotte Brøns, PhD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: H-4-2014-128
Record Dates: First submitted 2016-08-23; First posted 2016-12-05 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Type 2 Diabetes Mellitus; Insulin Resistance; Dyslipidemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance; Dyslipidemias | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low birth weight (LBW) (Experimental): 25 males born at term (weeks 39-41) in 1979-1981 with LBW (BW<10th percentile)
  Interventions: Dietary Supplement: High carbohydrate overfeeding; Behavioral: Exercise; Behavioral: Normal physical activity
- Normal birth weight (NBW) (Experimental): 25 BMI- and age-matched males born at term (weeks 39-41) with normal birth weight (NBW) control individuals (BW: 50-90th percentile)
  Interventions: Dietary Supplement: High carbohydrate overfeeding; Behavioral: Exercise; Behavioral: Normal physical activity

INTERVENTIONS:
Dietary Supplement: High carbohydrate overfeeding — All participant's individual energy requirement will be determined in mega joules (MJ) per day. The energy requirement will be multiplied by a factor 1.5 for a low physical activity level (PAL). The MJ will be rounded up or down to the nearest whole number.
  The participant will receive food corresponding to ~25% additional energy above their calculated energy requirement. The 25% extra energy will be supplied to the participants for 4 weeks in the form of food containing simple carbohydrates. The subjects will be given a daily snack package containing processed foods or refined foods such as sweets, cookies, soft drinks, juice etc. To ensure an adequate energy surplus (i.e. weight gain), physical activity has to be decreased to a low level during the 4 weeks overfeeding period.
Behavioral: Exercise — Half of the participants will be randomized to a 3-month exercise-training program.
  The training program consists of combined aerobic training and strength training. The training program is performed unsupervised 3 times per week 45 minutes per session for 3 months in the local fitness center. Before engaging in the training program a maximal oxygen consumption test (VO2 max) are conducted and the maximal heartrate (HR) are determined.Participants are wearing the Polar V800 HR monitor and are asked to note their HR in a training log at the end of the last interval at each training session. The strength training program consist of 6 exercises (2 exercises paired together) involving the large muscle groups. The first training session is completed supervised at Rigshospitalet . After 6 weeks the training program is adjusted. Compliance will be ensured by phone calls, text messages and e-mails from study personnel.
Behavioral: Normal physical activity — The other half of the participants will be randomized to a 3-month with normal physical activity level (control).
  The participants will have to return to the physical activity level they had before entering the study (baseline level). Compliance will be ensured by phone calls and text messages from study personnel. The subjects will wear a simple pedometer on the hip showing the number of steps. Once a week a text message (SMS-track) is automatically sent asking the participants to enter the weekly number of steps. The test personnel receive the reply and contact the participant if the number of steps does not match the baseline level. During the first and the last 7 days of the exercise intervention participants are wearing 2 accelerometers measuring their physical activity behavior.

SUMMARY:
Low birth weight (LBW), a marker of impaired fetal growth is an independent and strong risk factor for type 2 diabetes (T2D). A western lifestyle characterized by a surplus of calories, and/or a low physical activity level, associated with increased fat storage and altered lipid metabolism plays a central role in the pathogenesis of insulin resistance and T2D. Using state-of-the-art large-scale integrative physiology studies combined with basic studies of adipose and muscle tissue stem cell functions, the investigators aim to determine if LBW individuals exhibit decreased subcutaneous adipose tissue expandability, postprandial hyperlipidaemia and ectopic fat accumulation when exposed to 4 weeks of carbohydrate overfeeding. The investigators will subsequently examine if exercise training can revert and/or minimize the deleterious effects of carbohydrate overfeeding in a possibly birth weight differential manner.

ELIGIBILITY:
Inclusion Criteria:

* without known disease (approved health examination)
* caucasian
* born at term (weeks 39-41) in Denmark
* recruited from the national Danish Birth Registry
* born with either low or normal birthweight (see previous)

Exclusion Criteria:

* family history of diabetes in two generations (1st and 2nd degree relatives)
* self-reported high physical activity level (>10hrs /week).
* weight loss/gain >3 kg within the past 6 months
* alcohol intake of more than general recommendations
* substance abuser
* intake of medication know to affect outcomes

Ages: 35 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2016-08; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Adipose tissue expandability | baseline
  Percent (%) subcutaneous, visceral adipose tissue and hepatic fat will be determined by MR scanning in the two groups
Adipose tissue expandability | Difference between the two groups at baseline, after 4 weeks overfeeding and after 12 weeks exercise training.
  Percent (%) subcutaneous, visceral adipose tissue and hepatic fat will be determined by MR scanning in the two groups

SECONDARY OUTCOMES:
Glucose turnover rate | Baseline, 4 weeks overfeeding, 12 weeks training
  Turnover rates will be measured after a 5 hr mealtest by use isotopic tracers in the two groups
Lipid turnover rate | Baseline, 4 weeks overfeeding, 12 weeks training
  Turnover rates will be measured after a 5 hr mealtest by use isotopic tracers in the two groups
Epigenetics | Baseline, 4 weeks overfeeding, 12 weeks training
  Marks of adipose tissue, skeletal muscle stem cell and differentiated cell type genomes.

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Brøns, PhD, Principal Investigator — Rigshospitalet, Denmark; Allan Vaag, PhD, DMsc, Study Director — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Denmark, Copenhagen, Capital Region, Denmark